CLINICAL TRIAL: NCT04237623
Title: Phase II Trial Evaluating the Efficacy and Safety of Sargramostim Post-Infusion of T-Replete HLA Mismatched Peripheral Blood Haploidentical Hematopoietic Stem Cells and With Post Transplant Cyclophosphamide
Brief Title: GM-CSF With Post-Transplant Cyclophosphamide
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northside Hospital, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NSH 1246
Record Dates: First submitted 2020-01-17; First posted 2020-01-23 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Transplant-Related Hematologic Malignancy
MeSH Terms: interventions — sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GM-CSF post-transplant (Experimental): Sargramostim (GM-CSF) will start on Day +5 and continue until ANC >1000 x3 days or >1500 x1 day. GM-CSF will be administered not less than 24 hours after the last dose of cyclophosphamide and will be given at a dose of 250mcg/m2/day as an infusion over 2 hours.
  Interventions: Drug: Sargramostim; Other: Control Arm

INTERVENTIONS:
Drug: Sargramostim — 250mcg/m2/day IV starting Day +5
  Other Names: GM-CSF
Other: Control Arm — Standard G-CSF given to those who decline to receive GM-CSF
  Other Names: G-CSF

SUMMARY:
Given the increased number of HLA-mismatched haploidentical transplantation with post-transplant cyclophosphamide performed each year and the high risk of infectious complications associated with this type of transplant, the investigators suggest that GM-CSF administration post-infusion of T-replete haploidentical stem cells and post-transplant cyclophosphamide can yield similar count recovery rates to G-CSF with a potential of lowering risk of infectious complications.

ELIGIBILITY:
Inclusion Criteria:

* Availability of 5/10 to 8/10 matched related donor
* KPS >/= 70%
* CML, AML, MDS, ALL, CLL, HD, NHL, MPS/CMML, MM, any other hematologic condition deemed an eligible indication for allogeneic transplant by the treating center

Exclusion Criteria:

* Poor cardiac, pulmonary, liver, and renal function
* HIV-positive
* Patients who have a debilitating medical or psychiatric illness that would preclude them from giving informed consent
* History of severe or serious allergic reaction to human GM-CSF or yeast-derived products

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2020-05-18 (Actual); Primary Completion 2026-09-18 (Estimated); Study Completion 2026-09-18 (Estimated)

PRIMARY OUTCOMES:
The number of patients who achieved neutrophil engraftment at 20 days after the initiation of treatment. | 3 months after initial treatment
  The aim of the study is to establish equivalent effectiveness of Sargramostim to a matched control cohort of G-CSF treated patients in time to achieve neutrophil (ANC >500 x3 days) post infusion of HLA-mismatched peripheral blood haploidentical stem cells with post-transplant cyclophosphamide. Patients will be followed for 3 months following the initiation of treatment to see engraftment numbers at 20 days after initial treatment.

SECONDARY OUTCOMES:
How many patients are still alive measured by overall survival at 12 months following the initiation of treatment. | 12 months following initiation of treatment
  To estimate overall survival
How many patients have not relapsed measured by relapse rates at 12 months following the initiation of treatment. | 12 months following initiation of treatment
  To estimate relapse rates
How many patients develop graft-versus-host-disease (GVHD) measured by the incidence of GVHD at 12 months following initiation of treatment | 12 months following initiation of treatment
  To estimate incidence of GVHD
How many patients have not relapsed measured by progression-free survival at 12 months following the initiation of treatment | 12 months following initiation of treatment
  To estimate non-relapse mortality
How many patients died due to infections measured by the incidence and type of infections at 12 months following initiation of treatment | 12 months following initiation of treatment
  To estimate infection-related mortality
How many patients died due to a treatment-related adverse events grade 2 or greater as assessed by CTCAE v.4.0 | 12 months following initiation of treatment
  To estimate event-free survival
Number of patients to achieve full donor chimerisms at Days 30, 50, 100, and 6 months post-transplant as measured by donor chimerism data | 12 months following initiation of treatment
  To estimate graft failure
Number of patients that acquired an infection in the first 100-days post-transplant as measured by the incidence of infections | 12 months following initiation of treatment
  To estimate the rate of infections
Number of patients achieving platelet engraftment as measured by platelets reaching 20,000 without transfusion for 7 days | 12 months following initiation of treatment
  To assess time to platelet engraftment

CONTACTS AND LOCATIONS:
Overall Officials: Melhem Solh, MD, Principal Investigator — Northside Hospital
Locations (1):
- Northside Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No